CLINICAL TRIAL: NCT06543095
Title: Rib Removal in Retroperitoneal Open Partial Nephrectomy: Not As Painful As It Seems
Brief Title: Rib Removal and Pain in Partial Nephrectomy
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gokhan Sonmez, Assoc. Prof., TC Erciyes University
Other Study IDs: 2022/589
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pain; Partial Nephrectomy; Kidney Cancer
Keywords: Rib Removal; Partial nephrectomy; pain; renal cancer
MeSH Terms: conditions — Pain; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: who underwent rib removal during the partial nephrectomy
  Interventions: Other: Pain level
- Group 2: who didn't underwent rib removal during the partial nephrectomy
  Interventions: Other: Pain level

INTERVENTIONS:
Other: Pain level — Post-operative pain levels of the patients with detected using VAS score.

SUMMARY:
In this study, the effect of rib removal on postoperative pain in kidney cancer patients undergoing retroperitoneal open partial nephrectomy with flank incision was investigated. For this purpose, VAS score surveys were prepared for patients who underwent partial nephrectomy surgery in the early and late postoperative periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years who underwent open renal surgery due to kidney cancer were included in the study.

Exclusion Criteria:

* Patients with a preoperative (one day before surgery) VAS score greater than 0,
* Those with additional known diseases that could cause pain (herniated disc, urinary stone disease, inflammatory bowel diseases, other intra-abdominal pathologies),
* Intraoperative complications that could cause postoperative pain, metastasis, positive surgical margins or peri-renal invasion,
* Those who underwent laparoscopic surgery or those who converted to open surgery after laparoscopic surgery,
* Patients that regularly used painkillers for other reasons,
* Patients whose ribs other than the 11th rib were removed were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent open partial nephrectomy with flank incision between July 2022 and October 2023 in our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Pain level | days 0, 1, and 3 and week 3
  Primary outcome of the study was to compare the pain intensities of the two groups at postoperative days 0, 1, and 3 and week 3 and to evaluate the additional pain burden induced by the rib removal procedure.

SECONDARY OUTCOMES:
Complications | Postoperative 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data available on request from the authors